CLINICAL TRIAL: NCT05733585
Title: "A Physician-initiated, Observational, Prospective, Monocentric Study of Patients Treated With PuraBond Haemostatic Agent During Abdominal Aorta Open Repair "- PuraBond Study
Brief Title: Clinical Study of Patients Treated With PuraBond Haemostatic Agent During Abdominal Aorta Open Repair
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Mascia Daniele, Principal Investigator, IRCCS San Raffaele
Other Study IDs: PuraBond Study
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Hemostatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with abdominal aortic pathology: Patients with abdominal aortic pathology (aneurysmal or steno occlusive disease) candidate to open repair with PuraBond haemostatic agent.
  Interventions: Device: Purabond

INTERVENTIONS:
Device: Purabond — hemostatic efficacy of PuraBond

SUMMARY:
Purabond Study is a physician-initiated, observational, monocentric prospective Trial.

The aim of the study is to investigate the hemostatic efficacy of PuraBond for aortic anastomoses and suture lines in patients with abdominal aortic pathology (aneurysmal or steno occlusive disease) candidate to open repair at Vascular Surgery Departement - San Raffaele Hospital (Milan, Italy). The Study will include 100 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ≥ 18 years of age, presenting with an abdominal aortic aneurysm (pararenal, juxtarenal, infrarenal, aorto-iliac mono/bilateral)
* Use of the Purabond hemostatic agent in patients who, in the opinion of the Physician, don't have a satisfactory surgical haemostasis
* Patients ≥ 18 years of age with steno-occlusive abdominal aortic or iliac disease
* Patients that will treated by open repair , encompassing elective, urgent and emergency presentation, hospitalized and enrolled in Vascular Surgery Unit, San Raffaele Hospital (Milan, Italy)
* Patients able to sign specific informed consent for the study

Exclusion Criteria:

* Patients whom exhibited preoperative derangements in haematological and coagulation profiles, and baseline derangements in liver function
* Patients with abdominal aortic and/or iliac arteries disease candidate for endovascular treatment
* Pregnant, breastfeeding, or planning on becoming pregnant within 24 months
* Systemic infection (for example: sepsis)
* Impossibility or refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Study will include 100 patients with abdominal aortic pathology (aneurysmal or steno occlusive disease) candidate to open repair with PuraBond haemostatic agent in Vascular Surgery Unit, San Raffaele Hospital (Milan, Italy)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Time to Hemostasis | during the surgery
  time that goes from declamping to closing the abdomen

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berger JS, Hochman J, Lobach I, Adelman MA, Riles TS, Rockman CB. Modifiable risk factor burden and the prevalence of peripheral artery disease in different vascular territories. J Vasc Surg. 2013 Sep;58(3):673-81.e1. doi: 10.1016/j.jvs.2013.01.053. Epub 2013 May 2. PMID 23642926
- [Background] Diehm C, Schuster A, Allenberg JR, Darius H, Haberl R, Lange S, Pittrow D, von Stritzky B, Tepohl G, Trampisch HJ. High prevalence of peripheral arterial disease and co-morbidity in 6880 primary care patients: cross-sectional study. Atherosclerosis. 2004 Jan;172(1):95-105. doi: 10.1016/s0021-9150(03)00204-1. PMID 14709362
- [Background] Shander A, Kaplan LJ, Harris MT, Gross I, Nagarsheth NP, Nemeth J, Ozawa S, Riley JB, Ashton M, Ferraris VA. Topical hemostatic therapy in surgery: bridging the knowledge and practice gap. J Am Coll Surg. 2014 Sep;219(3):570-9.e4. doi: 10.1016/j.jamcollsurg.2014.03.061. Epub 2014 Jun 2. No abstract available. PMID 25151345